CLINICAL TRIAL: NCT06502769
Title: Efficacy of Therapeutic Exercise and Pain Neurophysiology Education in Temporomandibular Disorders: a Single-blind Randomized Controlled Trial
Brief Title: Efficacy of Therapeutic Exercise and Pain Neurophysiology Education in Temporomandibular Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, María Teresa Ortiz Moreno, MSc, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Temporomandibular Disorders
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Temporomandibular Disorder
Keywords: therapeutic exercise; pain neurophysiology; temporomandibular disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TE+PNE group (Experimental): patients with TMD who are going to combine therapeutic exercise with education in pain neurophysiology
  Interventions: Behavioral: Therapeutic Exercise; Behavioral: Pain Neurophysiology Education
- TE group (Other): patients with TMD who are going to perform isolated therapeutic exercise
  Interventions: Behavioral: Therapeutic Exercise

INTERVENTIONS:
Behavioral: Therapeutic Exercise — A therapeutic exercise program will be carried out
Behavioral: Pain Neurophysiology Education — A PNE program will be carried out
  Arms: TE+PNE group

SUMMARY:
The aim of this study is to compare the effects in pain of two different treatments in pacients with temporomandibular disorders (TMD). One group will receive isolated therapeutic exercise (TE) and the other will receive TE combined with pain neurophysiology education (PNE). The hypothesis of this study is that the PNE+TE group will obtain superior therapeutic results than an isolated TE program.

DETAILED DESCRIPTION:
Objective: To evaluate the differences in pain intensity by performing isolated therapeutic exercise (TE) versus performing the same exercise combined with pain neurophysiology education (PNE) in patients with temporomandibular disorders (TMD).

Design: Single-blind randomized controlled trial. Setting: Faculty of Physical Therapy of Alcalá de Henares. Participants: Subjects with TMD lasting more than 6 months (N= 36). Interventions: Participants will be randomly assigned to receive a TE program consisting of stretching, coordination and strengthening exercises (n= 18) or the same TE program in addition to a PNE program (n= 18), performed in two sessions of 40 minutes in groups of 6 participants. The intervention will last 12 weeks, where all participants must complete the exercise program daily, one year later they will be evaluated again.

Main outcome measures: The primary outcome will be pain intensity through the visual analogue scale (VAS) which will be completed at baseline, immediately after treatment, at 4 and 12 weeks and one year after treatment. Secondary outcome measures include pain-free mouth opening, Craniofacial Pain and Disability Inventory (CF-PDI), Pain Catastrophizing Scale (PCS), Tampa Scale for Kinesiophobia for Temporomandibular Disorders (TSK-11), pressure pain thresholds (PPT) and Patient Global Impression of Change (PGIC). They will be recorded through blinded assessments performed by 2 physiotherapists at baseline, immediately after treatment, 4 and 12 weeks after treatment. Student's t test will be used to determine differences between group interventions.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Limitation of mouth opening and/or jaw pain lasting more than 6 months
* Being able to understand the objective and carry out the study procedures
* Sign the informed consent.

Exclusion Criteria:

* Suffer from any underlying disease
* Pain due to tumors or infections, metastases, osteoporosis, inflammatory arthritis or fractures
* Be receiving any other treatment for TMD or consuming some type of substance that alters muscle tone.
* Patients with myopathies, diseases of the Peripheral Nervous System, mental disorders diagnosed by a doctor
* Inability to collaborate
* Any other situation in which the evaluation could be altered.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | The scale will be passed at baseline, immediately after treatment, at 4 and 12 weeks and one year after treatment.
  The intensity of pain will be evaluated using the Visual Analogue Scale that is represented by a 10cm line where the left end indicates "no pain" and the right end indicates "maximum pain".

SECONDARY OUTCOMES:
Mouth opening without pain | at baseline, immediately after treatment, 4 and 12 weeks after treatment.
  The distance between the upper and lower mandibular central incisors will be measured using a TheraBite range of motion scale.
Orofacial disability and pain | at baseline, immediately after treatment, 4 and 12 weeks after treatment.
  The CF-PDI is a self-administered questionnaire that measures pain and disability outcomes related to craniofacial pain. It consists of 21 items, with a score ranging from 0 to 63 points. A higher score reflects higher levels of disability.
Catastrophism | at baseline, immediately after treatment, 4 and 12 weeks after treatment.
  The PCS consists of a self-administered questionnaire with 13 items for the evaluation of catastrophic thoughts. It is divided into three domains: helplessness, magnification and rumination. Higher values denote greater pain catastrophizing
Kinesiophobia | at baseline, immediately after treatment, 4 and 12 weeks after treatment.
  The Spanish version of the TSK-11 will be used to evaluate the fear of re-injury due to movement. This questionnaire has a structure of 11 items and 2 factors that includes avoidance and harm of activities. Higher scores reflect greater fear of movement
Pressure pain thresholds | at baseline, immediately after treatment, 4 and 12 weeks after treatment.
  The masseter and anterior temporal PPTs will be assessed bilaterally using an analog algometer. Measurements will be reported in kg/cm2. The points will always be evaluated in the same order and will be repeated three times, with an interval of 1 minute. For each point the average of the three measurements will be considered.
Self-Perception of Improvement | at baseline, immediately after treatment, 4 and 12 weeks after treatment.
  PGIC will be used to assess perceived improvement after treatment (range, 0-7). Higher scores will indicate greater improvement

CONTACTS AND LOCATIONS:
Overall Officials: María Teresa Ortiz-Moreno, MSc, Principal Investigator — University of Alcalá; Gema Bodes-Pardo, PhD, Study Director — University of Alcalá
Locations (1):
- Campus Científico Tecnológico UAH. AV. de León, 3A., Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calixtre LB, Gruninger BL, Haik MN, Alburquerque-Sendin F, Oliveira AB. Effects of cervical mobilization and exercise on pain, movement and function in subjects with temporomandibular disorders: a single group pre-post test. J Appl Oral Sci. 2016 May-Jun;24(3):188-97. doi: 10.1590/1678-775720150240. PMID 27383698
- [Background] Chellappa D, Thirupathy M. Comparative efficacy of low-Level laser and TENS in the symptomatic relief of temporomandibular joint disorders: A randomized clinical trial. Indian J Dent Res. 2020 Jan-Feb;31(1):42-47. doi: 10.4103/ijdr.IJDR_735_18. PMID 32246680
- [Background] Sousa BM, Lopez-Valverde N, Lopez-Valverde A, Caramelo F, Fraile JF, Payo JH, Rodrigues MJ. Different Treatments in Patients with Temporomandibular Joint Disorders: A Comparative Randomized Study. Medicina (Kaunas). 2020 Mar 5;56(3):113. doi: 10.3390/medicina56030113. PMID 32151101
- [Background] Dos Santos Aguiar A, Bataglion C, Felicio LR, Azevedo B, Chaves TC. Additional effect of pain neuroscience education to craniocervical manual therapy and exercises for pain intensity and disability in temporomandibular disorders: a study protocol for a randomized controlled trial. Trials. 2021 Sep 6;22(1):596. doi: 10.1186/s13063-021-05532-x. PMID 34488856
- [Background] Wanman A, Marklund S. Treatment outcome of supervised exercise, home exercise and bite splint therapy, respectively, in patients with symptomatic disc displacement with reduction: A randomised clinical trial. J Oral Rehabil. 2020 Feb;47(2):143-149. doi: 10.1111/joor.12888. Epub 2019 Sep 30. PMID 31520538
- [Background] Yamaguchi Y, Sakuma S, Takagi S, Ogi N, Kurita K, Ariji Y, Taguchi N. Efficacy of therapeutic exercise for temporomandibular disorders as assessed by magnetic resonance imaging: a case report. J Phys Ther Sci. 2020 Jul;32(7):477-482. doi: 10.1589/jpts.32.477. Epub 2020 Jul 3. PMID 32753791
- [Background] Garrigos-Pedron M, La Touche R, Navarro-Desentre P, Gracia-Naya M, Segura-Orti E. Effects of a Physical Therapy Protocol in Patients with Chronic Migraine and Temporomandibular Disorders: A Randomized, Single-Blinded, Clinical Trial. J Oral Facial Pain Headache. 2018 Spring;32(2):137-150. doi: 10.11607/ofph.1912. PMID 29694464
- [Background] Michelotti A, de Wijer A, Steenks M, Farella M. Home-exercise regimes for the management of non-specific temporomandibular disorders. J Oral Rehabil. 2005 Nov;32(11):779-85. doi: 10.1111/j.1365-2842.2005.01513.x. PMID 16202040
- [Background] Malfliet A, Kregel J, Coppieters I, De Pauw R, Meeus M, Roussel N, Cagnie B, Danneels L, Nijs J. Effect of Pain Neuroscience Education Combined With Cognition-Targeted Motor Control Training on Chronic Spinal Pain: A Randomized Clinical Trial. JAMA Neurol. 2018 Jul 1;75(7):808-817. doi: 10.1001/jamaneurol.2018.0492. PMID 29710099
- [Background] Bodes Pardo G, Lluch Girbes E, Roussel NA, Gallego Izquierdo T, Jimenez Penick V, Pecos Martin D. Pain Neurophysiology Education and Therapeutic Exercise for Patients With Chronic Low Back Pain: A Single-Blind Randomized Controlled Trial. Arch Phys Med Rehabil. 2018 Feb;99(2):338-347. doi: 10.1016/j.apmr.2017.10.016. Epub 2017 Nov 11. PMID 29138049